CLINICAL TRIAL: NCT00042874
Title: An Open-Labeled, Non-Randomized Phase I Study of Alvocidib (Flavopiridol) Administered With Irinotecan (CPT-11) and Fluorouracil/Leucovorin in Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01410; 5757; NCI-5757; CDR0000069479; MSKCC-02024; U01CA069856 (NIH)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib; Irinotecan; Fluorouracil; Leucovorin

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes followed 5 hours later by leucovorin calcium IV over 2 hours and alvocidib IV over 1 hour immediately followed by 5-FU IV continuously over 48 hours beginning on day 1 of weeks 1, 3, and 5. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of alvocidib and 5-FU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Ten additional patients are treated at the MTD.
  Interventions: Drug: alvocidib; Drug: irinotecan hydrochloride; Drug: fluorouracil; Drug: leucovorin calcium; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. This phase I trial is studying the side effects and best dose of combination chemotherapy in treating patients with locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of flavopiridol (alvocidib) when administered with irinotecan hydrochloride, fluorouracil, and leucovorin calcium in patients with locally advanced or metastatic solid tumors.

II. Determine the clinical pharmacokinetics of fluorouracil when administered in this regimen in these patients.

III. Determine, preliminarily, the therapeutic activity of this regimen in these patients.Correlate the role of p21 and Drg1 with apoptosis and treatment response in patients receiving this regimen.

OUTLINE: This is a dose-escalation study of alvocidib and fluorouracil (5-FU).

Patients receive irinotecan hydrochloride IV over 90 minutes followed 5 hours later by leucovorin calcium IV over 2 hours and alvocidib IV over 1 hour immediately followed by 5-FU IV continuously over 48 hours beginning on day 1 of weeks 1, 3, and 5. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of alvocidib and 5-FU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Ten additional patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 27-77 patients will be accrued for this study within 11-38 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumor

  * Refractory to standard therapy or for which there is no standard therapy
  * Preference given to colorectal cancer, upper gastrointestinal cancer, or neuroendocrine tumors
* Evaluable disease
* No CNS metastases or primary CNS malignancy
* Performance status - Karnofsky 60-100%
* WBC at least 3,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Creatinine no greater than 1.5 mg/dL
* No history of cardiac arrhythmia
* No congestive heart failure
* No myocardial infarction within the past 6 months
* No prior grade 3 or 4 diarrhea secondary to irinotecan, despite optimal antidiarrheal prophylaxis
* HIV negative
* No serious or uncontrolled infection
* No other medical condition or reason that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 months after study participation
* At least 2 weeks since prior immunotherapy
* No more than 2 prior chemotherapy regimens unless there is no evidence of significant myelotoxicity as determined by the primary investigator
* At least 2 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin)
* Prior irinotecan and fluorouracil allowed
* At least 2 weeks since prior radiotherapy
* Recovered from all prior therapy
* No other concurrent investigational medications
* No concurrent vitamins, antioxidants, or herbal preparations or supplements except a single daily multivitamin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2002-05; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
MTD of biweekly flavopiridol when given in conjunction with irinotecan hydrochloride, fluorouracil, and leucovorin | 8 weeks

SECONDARY OUTCOMES:
Clinical pharmacokinetics of the regimen under investigation | Day 1, prior to flavopiridol infusion (t=3:30hr), post flavopiridol infusion (t=4:30hr), prior to flavopiridol infusion (t=3:30hr), post 30 minute flavopiridol bolus (t=4:00), post 4 hour flavopiridol infusion (t=8:00hr)
Therapeutic activity of flavopiridol in combination with irinotecan hydrochloride in patients with advanced solid tumors | Up to 7 years
Change in molecular marker expression | Baseline to 2 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States